CLINICAL TRIAL: NCT05154006
Title: Promoting Self-efficacy and Social Support to Enable Women to Reduce the Risks of Pelvic Organ Prolapse Related to Heavy Lifting in a Non-randomized Controlled Trial With a 3-arm Parallel Intervention Group Design in Rural Nepal
Brief Title: Women Lift Safely! An Intervention Study to Reduce the Risks of Heavy Lifting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Suzanne und Hans Biäsch Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 41487
Record Dates: First submitted 2021-12-09; First posted 2021-12-10 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Behavior, Health; Behavior, Maternal; Work Related Stress
Keywords: Pelvic organ prolapse; Self-efficacy; Social support; Health behavior change
MeSH Terms: conditions — Health Behavior; Behavior; Occupational Stress; Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: 3-arm parallel non-randomized controlled trial
Who Masked: Participant
Masking Description: The assignment of groups to the villages will be random (drawing lots by a person not included in the research team). All participants from one village will receive the same intervention. Participants are blinded to condition. Enumerators cannot be blinded to condition, but the specific intervention assignment is concealed until the arrival at the intervention site. In a debriefing after the follow up interviews, the allocated intervention group will be revealed to the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Control (Information only) (Active Comparator): Women in the active control group receive instruction on safe carrying behaviors (reduce carried weight & use safe lifting techniques) and information about benefits when performing the behavior and reducing strain on the pelvic floor.
  Interventions: Behavioral: Information about benefits of the behavior; Behavioral: Instruction on how to perform a behavior
- Individual promotion of self-efficacy (Experimental): The group "Individual promotion of self-efficacy" receives the same instructions and information on safe carrying behavior as the control group.
  Additionally, this group will receive behavior change techniques (Michie et al., 2013) to increase self-efficacy (psychological activities to increase self-confidence / belief in own capability to reduce risks of carrying loads with own behavior).
  Interventions: Behavioral: Information about benefits of the behavior; Behavioral: Instruction on how to perform a behavior; Behavioral: Self-efficacy
- Promotion of self-efficacy + social support (Experimental): The group "Promotion of self-efficacy + social support" receives the same instructions for safe carrying behavior as the control group. The intervention will also include the same behavior change techniques to promote self-efficacy.
  Additionally, a social partner from the same or neighboring household will be involved in the intervention activities. The partner will participate in the intervention activities and will be instructed to provide emotional, practical and informational social support.
  Interventions: Behavioral: Information about benefits of the behavior; Behavioral: Instruction on how to perform a behavior; Behavioral: Self-efficacy; Behavioral: Social Support

INTERVENTIONS:
Behavioral: Information about benefits of the behavior — The women will be informed that the safe carrying behaviors can reduce pelvic strain. She is informed about the benefits reducing pelvic strain may imply [5.1; 5.3.,5.6 Information about health; environmental; social; and emotional consequences, (Michie et al., 2013)]
Behavioral: Instruction on how to perform a behavior — For the target behavior "reduce carried weight" information on recommended weight limits will be given. The women will be encouraged, that even if these limits may not be feasible for them, any reduction of weight can still reduce the strain on the pelvic floor.
  For the target behavior "safe lifting techniques", instructions to learn the correct behavior (how to perform safe lifting techniques?) based on leaflets developed and validated by Caagbay et al., (2017, 2020) [4.1 Instruction on how to perform a behavior (Michie et al., 2013)]
Behavioral: Self-efficacy — Self-efficacy will be promoted by the four sources of self-efficacy (Bandura, 1977): 1) Mastery Experiences (experience that one is able to successfully apply the behavior), vicarious experience (observing successful others performing the safe carrying behavior), verbal persuasion (receiving positive feedback when performing the behavior and encouraging messages to do so) and emotional state (e.g. being in a positive emotional state when performing the behavior). [6.1 Demonstration of the behavior; 8.1 Behavioral practice/rehearsal; 15.1 Verbal persuasion about capability; 15.2 Mental rehearsal of successful performance; 15.3 Focus on past success;15.4 Self-talk; 5.4 Monitoring of emotional consequences (Michie et al., 2013)]
  Arms: Individual promotion of self-efficacy; Promotion of self-efficacy + social support
Behavioral: Social Support — A self-selected social partner from the same or neighboring household (e.g. husband, mother-in-law) will be involved in the learning process (observational learning, feedback). The partner will participate in the intervention activities and will be instructed to provide emotional social support and practical informational support. [3.2 practical support, 3.3 emotional support; 6.3 Information about others' approval (Michie et al., 2013).]
  Arms: Promotion of self-efficacy + social support

SUMMARY:
The Women Lift Safely! Intervention study aims to increase safe carrying behavior to reduce health risks of heavy lifting in a rural area of Nepal (i.e. reducing weight and using safe lifting techniques).

The study's specific aims are to:

1) Test whether a psychological intervention that promotes self-efficacy can promote women's use of safe carrying behavior effectively compared to an information only control condition.

(2) Test whether including a social partner in the intervention is more effective than an individual psychological intervention.

DETAILED DESCRIPTION:
Background

The frequent carrying of heavy loads bears health risks for women in low- and middle-income countries, such as Nepal (Geere et al. 2018,2020; Koyucu et al., 2021; Walker & Gunasekera, 2011).

To prevent the physical health impacts of carrying heavy loads, e.g. pelvic organ prolapse, research has shown that preventive behaviors in terms of applying safe carrying behaviors can enable women to minimize adverse health outcomes:

1. Reducing the carried load, especially during pregnancy and postpartum (Darshan, 2009; Koyucu et al., 2021; MacDonald et al., 2013; Oxford University Hospitals, 2016; Sharma, 2012; SUVA, the Swiss National Accident Insurance Fund, 2019)
2. Using safe lifting techniques (exhale, tighten pelvic floor and use a safe body posture when lifting load) (Caagbay et al., 2020; Hagins et al., 2004)

In a preliminary study, the investigators identified low self-efficacy (belief in the own capability to engage in healthy behavior) and insufficient social support (emotional, practical or informational assistance by social partner) as reasons for risky carrying behavior (Tomberge et al., 2021).

Study design

A 3-arm parallel non-randomized controlled trial will be conducted in three rural villages in the Kavre and Sindhupalanchowk districts of Nepal. The villages will be randomly assigned to one of the three groups: (1) individual promotion of self-efficacy, (2) promotion of self-efficacy + social support (3) active control group to test the effect of promoting self-efficacy and the additional effect of social support on safe carrying behavior against an information only control group. The latter, in the sense of a waiting list control group, will receive the most effective intervention after completing the study. The assignment of groups to the villages will be random (drawing lots by a person not included in the research team). All participants from one village will receive the same intervention. This village-based allocation of interventions prevents the transfer of information within the village (spillover effect, Benjamin-Chung et al., 2018).

Recruitment and informed consent procedure:

The villages included were already part of the prestudy in 2019. 100 women from each of the three villages and a self-selected social partner from the same or neighboring household (e.g. husband, mother-in-law) having experience in carrying loads will be included (N = 600). Households / Participants within the villages will be selected using the random route method (Hoffmeyer-Zlotnik, 2003). Due to their acute vulnerability, women who are pregnant or who have delivered in the last month will be approached specifically.

Arriving at the households, trained local research assistants will present themselves and briefly inform about the study purpose and procedures in Nepali language. The respondents willing to participate will be provided with more detailed explanation of the study both verbally and with participant information sheets. Respondents will also be provided with information and consent forms written in easy language and will be informed that the participation will be voluntary.

Since all the participants will be interviewed in personal communication with enumerators with a professional background in health science the informed consent will be fully read out to the participants and can be explained more deeply in case of any dubiety. After explaining the content of the study the participant will ask the woman if she and also a self-selected social partner are willing to participate in the study. If the women and the social partner agree and all their doubts and questions are answered, they will be requested to sign the informed consent sheet either by signature or thumbprint.

Study procedure:

Training: Before the beginning of the study, the local team (practitioners graduated in nursing sciences or physiotherapy and research assistants graduated in health/social Sciences) will be trained in interviewing techniques and data collection tools. Additionally, a pelvic physiotherapist will train them in instructing and assessing safe lifting techniques.

The training will last one week, 2 pretests in villages not part of the analyses included.

Baseline Survey and Intervention:

The research assistants will conduct baseline interviews in one village. They will collect quantitative data in computer-assisted, structured face-to-face interviews with women and their social partners and conduct structured behavioral observations of the women while carrying a water-filled container. A local field coordinator will monitor the quality of data during the data collection during fieldwork to reduce interviewer bias.

After the baseline interview, the households will be visited again by the health practitioners in order to receive one of the three interventions to promote safe carrying behaviors (information only control, individual promotion of self-efficacy, promotion of self-efficacy + social support) for which the study participants will be blinded. The study team cannot be blinded to condition, but the specific intervention assignment is concealed until the arrival at the intervention site. The intervention will be delivered via household visits.

Follow-Up:

The follow-up survey to test intervention effects will be conducted 8 weeks after baseline. In a debriefing after the follow up survey, the allocated intervention group will be revealed to the participants.

Hypotheses:

The main research questions and hypotheses of this study are:

1. Does the promotion of self-efficacy lead to more safe carrying behavior in women?

   H1a: Women in the two intervention groups with self-efficacy promotion indicate increased reduction of carried weight compared to the control group.

   H1b: Women in the two intervention groups with self-efficacy promotion indicate increased use of safe lifting techniques compared to the control group.
2. Can adding social support by a social partner increase safe carrying behavior additionally?

   H2a: Women in the group with self-efficacy + social support indicate increased reduction of carried weight compared to the group with individual self-efficacy promotion.

   H2b: Women in the group with self-efficacy + social support indicate increased use of safe lifting techniques compared to the group with individual self-efficacy promotion.
3. Can the intervention effects on safe carrying behavior be explained by increased self-efficacy?

   H3a: The intervention effect on carried weight of the two intervention groups with self-efficacy promotion compared to controls is explained by increased self-efficacy.

   H3b: The intervention effect on the use of safe lifting techniques in the two intervention groups with self-efficacy promotion compared to controls is explained by increased self-efficacy.

   H3c: The increased reduction of carried weight of the group self-efficacy + social support compared to the group with individual self-efficacy promotion is explained by increased self-efficacy.

   H3d: The increased use of safe lifting techniques in the group self-efficacy + social support compared to the group with individual self-efficacy promotion is explained by increased self-efficacy.
4. Can the intervention effects be explained by increased received social support? H4a: The increased reduction of carried weight of the group self-efficacy + social support compared to the group with individual self-efficacy promotion is explained by increased social support.

   H4b: The increased use of safe lifting techniques in the group self-efficacy + social support compared to the group with individual self-efficacy promotion is explained by increased social support.

   H4c: The increased self-efficacy in the group self-efficacy + social support compared to the group with individual self-efficacy promotion is explained by increased received social support.

   Additionally, the investigators will investigate the following exploratory research questions:
5. Can the interventions increase women's self-efficacy and intention to reduce carried weight in future pregnancies and postpartum?
6. Is the reduction of carried weight related to an increased carrying frequency?
7. Does the intervention have an impact on other psychosocial determinants of carrying behavior?
8. Can the interventions improve women's quality of life, and reduce strain during lifting, pain, symptoms of incontinence and pelvic organ prolapse, and perceived personal control over symptoms?
9. Do the interventions have an impact on relationship quality with the social partner and/ or the social partners' behavior and attitudes towards safe carrying behavior?

Statistics:

An a priori power analysis with a desired power of > 95%, a significance level of α = 0.05 and the assumption of medium effects (based on a study by Ernsting et al.,(2015)) resulted in a required sample size of N = 251 to detect a significant difference between the three groups when using repeated-measures ANCOVA (Faul et al., 2009). This analysis is based on including six covariates (Outcome at baseline, age, socioeconomic status, ethnicity, education and pregnancy status). Due to an expected dropout rate of up to 20% from baseline to follow-up (Wood et al., 2004) we will recruit 100 women in each of the three villages.

Planned analyses:

Summary of descriptive statistics

All primary and secondary outcomes will be presented. For the evaluation of the intervention effects, repeated measures covariance analyses (ANCOVA) with the two measurement points (pre/ post) will be calculated using the intervention groups as independent variables and reduced weight and use of safe lifting techniques as well as self-efficacy and social support as dependent variables. Further secondary outcomes, e.g. effects of the intervention on psychological wellbeing and physical health symptoms, will be calculated additionally.

Mediation analyses will be carried out for self-efficacy and social support as mediators.

Research Team:

Jennifer Inauen & Vica Tomberge (University of Bern, Institute of Psychology, Health Psychology and Behavioural Medicine), Akina Shrestha (Kathmandu University Hospital; Kathmandu University School of Medical Sciences), Regula Meierhofer (Eawag, Swiss Federal Institute of Aquatic Science and Technology; Department of Sanitation, Water and Solid Waste for Development), Helena Luginbühl (Bern University of Applied Sciences, Department of Health Professions, Division of Physiotherapy)

ELIGIBILITY:
Inclusion criteria:

* Written informed consent
* Gender: female
* Being adult and in reproductive age (18-49 years)
* Having experience in carrying loads
* Having a social partner with experience in carrying loads
* Residing in the targeted community

Exclusion criteria:

* If the women themselves or a household member presents covid symptoms they need to be excluded to avoid any risk of contamination of the research team.
* Women without a possible social partner will be excluded from the survey since this intervention is designed to include support of a social partner. They will receive the information only control intervention for ethical reasons when approached as a household in random selection.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Sex: Female
Enrollment: 600 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2022-04-02 (Actual); Study Completion 2022-10-22 (Actual)

PRIMARY OUTCOMES:
Self-reported carried weight at follow up | 8 weeks after intervention
  Carried weight will be assessed through the sum of two self-reported items referring to the weight carried in the last week. Open answers in kg.
  "In the last 7 days, what was the usual weight of water you carried per trip?" "In the last 7 days, what was the usual weight of other loads (e.g. grass, fodder, firewood you carried per trip?"
Index of self-reported safe lifting techniques during performance at follow up | 8 weeks after intervention
  An index of safe lifting will be calculated by the product of a safe lifting score x self-reported frequency of using safe-lifting techniques, ranging from 0 (= never uses safe lifting techniques) to 7 (= always uses safe lifting techniques)
  Score: The participants will be asked to lift a water-filled container at the size they usually carry. Lifting techniques will then be assessed through two self-reported items, e.g.:
  "What did you do with your pelvic floor during lifting?" 1 = "Tightening"; 0 "Relax"; 0 "did not feel the pelvic floor"; 0 = "I don't know"; 0 = "other".
  The safe lifting score is calculated by summing the points of the two items, thus ranging from 0 (= unsafe lifting) to 2 (= safe lifting).
  Frequency: Average of two items "In the last 7 days, how often did you tighten your pelvic floor when lifting loads?"; "In the last 7 days, how often did you exhale when lifting loads?" Answer options 1 = ((Almost) never (0%)) to 5 (= (Almost) always (100%)).

SECONDARY OUTCOMES:
Observed safe lifting techniques during performance | 8 weeks after intervention
  Local research assistants will conduct behavioral observations to examine lifting techniques.
  "Observe: Is she exhaling (breath) while lifting?" 1 ="yes"; 0 = "no". Answer option 1 refers to the safe lifting technique.
Self-reported perception and use of pelvic floor muscles during lifting through open questions | 8 weeks after intervention
  A secondary self-reported score assesses perception and use of pelvic floor muscles when lifting a water-filled container through two items with answering options coded 0 (= unsafe) or 1 (=safe) will serve to validate the answers given for the safe lifting score. The pelvic floor muscle score is calculated by summing the points:
  1. "Did you feel any muscles tightening during lifting?" "If yes, which ones?" 0 = "Back"; 0 = "Stomach";0 = "Legs"; 0 = "Head"; 0 = "Neck"; 0 = "Muscles of arms"; 1 ="Pelvic floor" "; 0 = "Other.
  2. "How did you tighten the pelvic floor muscles?" 1 = "Imagine stopping flow of urine"; 1 = "Feeling a lift inside the pelvis"; 1 = "Feeling a squeeze inside the pelvis"; 1 = "Small tightening of muscles in lower stomach"; 0 = "I don't know"; 1 = "other".
Self-reported self-efficacy to reduce carried weight | 8 weeks after intervention
  Average of self-reported five items based on the Health Action Process Approach (HAPA model; Schwarzer, 2008), e.g. "How sure are you that you can always reduce the carried load to your weight limit?" 1 = "not at all sure" to 5 = "very sure". Higher scores indicate stronger self-efficacy.
Self-reported self-efficacy to use safe lifting techniques | 8 weeks after intervention
  Average of five self-reported items based on the HAPA model (Schwarzer, 2008), e.g. "How sure are you that you are able to always use safe lifting techniques?" 1 = "not at all sure" to 5 = "very sure". Higher scores indicate stronger self-efficacy.
Self-reported received social support to reduce carried weight | 8 weeks after intervention
  Emotional, informational and instrumental support to reduce carried weight will be assessed self-reported by the Berlin Social Support Scale (Schwarzer & Schulz, 2013).
  Average of 9 items, e.g. "This person expressed concern about my decision to carry less weight." 1 = "not at all" to 5 = "very much". Higher scores indicate more social support.
Self-reported received social support to use safe lifting techniques | 8 weeks after intervention
  Berlin Social Support Scale (Schwarzer & Schulz, 2013). Average of 9 items, e.g. "This person encouraged me not to give up when trying to use safe lifting techniques." 1 = "not at all" to 5 = "very much". Higher scores indicate more social support.
Self-reported carrying frequency per week | 8 weeks after intervention
  Frequency will be calculated by the product of self-reported carrying trips "In the last 7 days, how many carrying trips did you conduct per day?" by days carried per week "On how many of the last 7 days did you carry loads?"
Self-reported self-efficacy to reduce carried weight during prospective pregnancies / postpartum | 8 weeks after intervention
  Average of three items, e.g. "How sure are you that you can always avoid to carry loads during and after pregnancy?" 1 = "not at all sure" to 5 = "very sure". Higher scores indicate stronger self-efficacy.
Self-reported weight intended to carry during prospective pregnancies / postpartum | 8 weeks after intervention
  3 self-reported items referring to intended carried weight per trip in the first half of pregnancy, the second half of pregnancy and three months postpartum, e.g. "In the first half of your pregnancy, what weight do you intend to carry per trip?" Answer in kg.
Self-reported risk perception to reduce carried weight | 8 weeks after intervention
  Average of two items based on the Health Action Process Approach (HAPA model; Schwarzer, 2008), e.g. "How high do you think the risk is that you get pelvic organ prolapse if you carried loads above the weight limit?" 1 = "not at all high" to 5 = "very high". Higher scores indicate higher risk perception.
Self-reported risk perception to use safe lifting techniques | 8 weeks after intervention
  Average of two items based on the HAPA model (Schwarzer, 2008), e.g. "How high do you think is the risk that you get pelvic organ prolapse if you do not use safe lifting techniques?" 1 = "not at all high" to 5 = "very high". Higher scores indicate higher risk perception.
Self-reported outcome expectancies to reduce carried weight | 8 weeks after intervention
  Average of two items based on the HAPA model (Schwarzer, 2008), e.g. "If I reduce the weight of the load I carry, I can protect myself from negative health impacts (e.g. pelvic organ prolapse)" 1 = "Agree not at all" to 5 = "agree very much". Higher scores indicate higher outcome expectancies.
Self-reported outcome expectancies to use safe lifting techniques | 8 weeks after intervention
  Average of two items based on the HAPA model (Schwarzer, 2008), e.g. "When using safe lifting techniques, I can protect myself from negative health impact (e.g. Pelvic organ prolapse)." 1 = "Agree not at all" to 5 = "agree very much". Higher scores indicate higher outcome expectancies.
Self-reported intention to reduce carried weight | 8 weeks after intervention
  Average of two items based on the HAPA model (Schwarzer, 2008), e.g. "How strongly do you intend to always reduce carried weight?" 1 = "not at all" to 5 = "very much". Higher scores indicate stronger intention.
Self-reported intention to use safe lifting techniques | 8 weeks after intervention
  Average of two items based on the HAPA model (Schwarzer, 2008), e.g. "How strongly do you intend to always use safe lifting techniques?" 1 = "not at all" to 5 = "very much". Higher scores indicate stronger intention.
Self-reported action planning to reduce carried weight | 8 weeks after intervention
  Action planning will be assessed based on the HAPA model (Schwarzer, 2008). The research assistant will ask "Have you made a detailed plan regarding… (1) "when to start", (2) "how", and (3) "how often" to reduce the weight of load carried?" The research assistant will code answers 1 (vs. 0) when a plan is mentioned.
Self-reported action planning to use safe lifting techniques | 8 weeks after intervention
  Action planning will be assessed based on the HAPA model (Schwarzer, 2008). The research assistant will ask "Have you made a detailed plan regarding… (1) "when to start", (2) "how", and (3) "how often" to use safe lifting techniques?" The research assistant will code answers 1 (vs. 0) when a plan is mentioned.
Self-reported coping planning to reduce carried weight | 8 weeks after intervention
  Coping planning will be assessed by one item based on the HAPA model (Schwarzer, 2008): "How can you overcome difficulties that prevent you from reducing the weight of load carried?". Answer options are precoded and coping planning will be rated dichotomous 1 (vs. 0) if any plan is mentioned.
Self-reported coping planning to use safe lifting techniques | 8 weeks after intervention
  Coping planning will be assessed by one item based on the HAPA model (Schwarzer, 2008): "How can you overcome difficulties that prevent you from using safe lifting techniques?". Answer options are precoded and coping planning will be rated dichotomous 1 (vs. 0) if any plan is mentioned
Self-reported perceived barriers to reduce carried weight | 8 weeks after intervention
  Perceived barriers will be assessed by one item based on the HAPA model (Schwarzer, 2008): "What do you think, how difficult would reducing carried weight be for you?" 1 = "not at all" to 5 = "very much".
Self-reported perceived barriers to use safe lifting techniques | 8 weeks after intervention
  Perceived barriers will be assessed by one item based on the HAPA model (Schwarzer, 2008): "What do you think, how difficult would using safe lifting techniques be for you?" 1 = "not at all" to 5 = "very much".
Additional self-reported psychosocial determinants to reduce carried weight | 8 weeks after intervention
  Determinants identified in a prestudy (Tomberge et al., 2021):
  Response efficacy: "Even if I reduce carried weight, I am not safe from getting pelvic organ prolapse." Spiritual beliefs: Two items, e.g. "Whether I get pelvic organ prolapse or not depends on gods' will rather than on my carrying behavior".
  Identity: Two items, e.g. "I would feel odd if I reduced the weight I usually carry. (reverse)" Affective attitudes: Two items, e.g. "How much do you like to carry a reduced weight when carrying loads?" Attitudes on the gender division of labor: Two items, e.g. "It is a woman's task exclusively to make sure all family members and livestock have enough food and water." Normative beliefs: Four items, e.g. "How much would people who are important to you approve if you reduced carried weight?".
  Decision making: Two items, e.g. "To what extent are you the only one to decide on how much weight you carry?" Answer options are 1 = e.g. "not at all" to 5 = e.g. "very much"
Additional self-reported psychosocial determinants of using safe lifting techniques. | 8 weeks after intervention
  Determinants identified in a prestudy (Tomberge et al., 2021):
  Response efficacy: "Even if I use safe lifting techniques, I am not safe from getting pelvic organ prolapse." Spiritual beliefs: Two items, e.g. "Whether I get pelvic organ prolapse or not depends on gods' will rather than on my carrying behavior".
  Identity: Two items, e.g. "Using safe lifting techniques is part of my identity/ who I am." Affective attitudes: Three items, e.g. "How much do you like to use safe lifting techniques?" Attitudes on the gender division of labor: Two items, e.g. "It is a woman's task exclusively to make sure all family members and livestock have enough food and water." Normative beliefs: Four items, e.g. "How much would people who are important to you approve if you used safe lifting techniques?".
  Decision making: Two items, e.g. "To what extent are you the only one to decide which techniques to use when you lift load?" Answer options are 1 = e.g. "not at all" to 5 = e.g. "very much"
Self-reported knowledge on safe carrying behaviors | 8 weeks after intervention
  Knowledge on how to carry loads in a safer way will be assessed through two self-reported items with answering options coded 0 (= correct) or 1 (= false). The safe lifting knowledge score is calculated by summing the points: "Can you tell me whether these are safe lifting techniques to reduce strain on the pelvic floor?" 0 = "Lift your toes up when lifting"; 1 = "Exhale (breath) when lifting"; 1 = "Reduce carried weight", 0 = "Use only one hand when lifting"; 0 = "Take a run-up before lifting"; 1 = "Tighten pelvic floor when lifting"; 0 = "Hold breath when lifting".
Self-reported knowledge on tightening pelvic floor | 8 weeks after intervention
  Knowledge on how to tighten the pelvic floor will be assessed through two self-reported items with answering options coded 0 (= correct) or 1 (= false). The pelvic floor knowledge score is calculated by summing the points: "Can you tell me whether the following are techniques to tighten the pelvic floor?" 1 = "Imagine to stop flow of urine"; 0 = "Bring shoulder blades together"; 1 = "Feeling a lift inside the pelvis"; 1 = "Small tightening of muscles in lower stomach"; 0 = "Bend knees"; 1 = "Lift toes up"; 0 = "Imagine to press as if going for defecation"; 1 = "Feeling a squeeze inside the pelvis".
Self-reported pain | 8 weeks after intervention
  Pain will be assessed by three items supported by the revised faces pain scale- (FPS-R) and the numerical pain rating scale (NPRS) (Pathak et al., 2018; Sharma et al., 2017) , e.g. "How much pain did you feel in your pelvis in the last 4 weeks?" 0 = "No pain" to 10 = "worst pain possible".
Self-reported strain during lifting | 8 weeks after intervention
  Strain during lifting will be assessed by two items right after lifting a water filled container, e.g. "How much strain did you feel in your pelvic floor when lifting the container?" 0 = "No strain at all" to 5= "very much strain". Higher scores indicate higher strain.
Self-reported symptoms of pelvic organ prolapse | 8 weeks after intervention
  Average of expression on seven self-reported symptoms (POP-SS; (Hagen et al., 2009)).
Self-reported symptoms of incontinence | 8 weeks after intervention
  Average of expression on five self-reported symptoms of incontinence will be assessed by a combination of selected items of the Incontinence Severity Index - 2 (ISI-2) and the Incontinence Symptom Index - Pediatric (ISI-P) (as used in (Parden et al., 2016)).
Self-reported quality of life | 8 weeks after intervention
  Average of eight items (EUROHIS-QOL 8-item index, (Rocha et al., 2012), e.g. "How satisfied are you with the conditions of your living place?" 1 = "not at all satisfied" to 5 = "very satisfied". Higher scores indicate higher quality of life.
Self-reported illness-related personal control | 8 weeks after intervention
  Average of six self-reported items (Personal control from the revised Illness Perception Questionnaire; Moss-Morris et al., 2002), e.g. "There is a lot which I can do to control my symptoms." 1 = "agree not at all" to 5 = "agree very much". Higher scores indicate higher illness-related personal control.
Self-reported daily functioning | 8 weeks after intervention
  One item "Please rate the severity by which carrying loads reduces your daily functioning." (Functioning rating scale; (de Jong et al., 2016)).
Self-reported quality of relationships | 8 weeks after intervention
  The quality of relationships between women and their social partners will be assessed by the average of seven self-reported items based on the Perceived Relationship Quality Components Inventory (PRQC, (Fletcher et al., 2000)); e.g. "How satisfied are you with your relationship with your social partner?" 1 = "not at all satisfied" to 5 = "very satisfied". Higher scores indicate improved relationship quality.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Inauen, PhD, Principal Investigator — University of Bern, Health Psychology & Behavioral Medicine; Akina Shrestha, PhD, Principal Investigator — Dhulikhel Hospital, Kathmandu University School of Medical Sciences
Locations (2):
- Nepal (2):
  - Outreach Centers of Dhulikhel Hospital, Kathmandu University School of Medical Sciences, Kavre, Kavre District
  - Outreach Centers of Dhulikhel Hospital, Kathmandu University School of Medical Sciences, Sindhupalchok

IPD SHARING:
Plan to Share IPD: Yes
Individual, anonymized participant data will be shared in the open science framework repository (OSF) after publishing the main outcomes of this study.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Study information and materials will be uploaded after the pretests. The Analysis Code and Participant data will be uploaded after the acceptance of a publication describing the main outcomes of the interventions.

REFERENCES:
- [Background] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061
- [Background] Benjamin-Chung J, Arnold BF, Berger D, Luby SP, Miguel E, Colford JM Jr, Hubbard AE. Spillover effects in epidemiology: parameters, study designs and methodological considerations. Int J Epidemiol. 2018 Feb 1;47(1):332-347. doi: 10.1093/ije/dyx201. PMID 29106568
- [Background] Caagbay D, Raynes-Greenow C, Dangal G, Mc Geechan K, Black KI. Impact of an informational flipchart on lifestyle advice for Nepali women with a pelvic organ prolapse: a randomized controlled trial. Int Urogynecol J. 2020 Jun;31(6):1223-1230. doi: 10.1007/s00192-020-04228-1. Epub 2020 Jan 31. PMID 32006071
- [Background] Caagbay DM, Black K, Dangal G, Raynes-Greenow C. Can a Leaflet with Brief Verbal Instruction Teach Nepali Women How to Correctly Contract Their Pelvic Floor Muscles? J Nepal Health Res Counc. 2017 Sep 8;15(2):105-109. doi: 10.3126/jnhrc.v15i2.18160. PMID 29016577
- [Background] Darshan, A. (2009). Prevalence of uterine prolapse amongst gynecology OPD patients in Tribhuvan university teaching hospital in Nepal and its sociocultural determinants. In Safe Motherhood Network Federation (SMNF), Beyond Beijing Committee (BBC). Tribhnuvan University Teaching Hospital (TUTH).
- [Background] de Jong K, Ariti C, van der Kam S, Mooren T, Shanks L, Pintaldi G, Kleber R. Monitoring and Evaluating Psychosocial Intervention Outcomes in Humanitarian Aid. PLoS One. 2016 Jun 17;11(6):e0157474. doi: 10.1371/journal.pone.0157474. eCollection 2016. PMID 27315263
- [Background] Ernsting A, Knoll N, Schneider M, Schwarzer R. The enabling effect of social support on vaccination uptake via self-efficacy and planning. Psychol Health Med. 2015;20(2):239-46. doi: 10.1080/13548506.2014.920957. Epub 2014 May 27. PMID 24862090
- [Background] Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G*Power 3.1: tests for correlation and regression analyses. Behav Res Methods. 2009 Nov;41(4):1149-60. doi: 10.3758/BRM.41.4.1149. PMID 19897823
- [Background] Fletcher, G. J. O., Simpson, J. A., & Thomas, G. (2000). The Measurement of Perceived Relationship Quality Components: A Confirmatory Factor Analytic Approach. Personality and Social Psychology Bulletin, 26(3), 340-354. https://doi.org/10.1177/0146167200265007
- [Background] Hagen S, Glazener C, Sinclair L, Stark D, Bugge C. Psychometric properties of the pelvic organ prolapse symptom score. BJOG. 2009 Jan;116(1):25-31. doi: 10.1111/j.1471-0528.2008.01903.x. Epub 2008 Oct 8. PMID 18947342
- [Background] Hagins M, Pietrek M, Sheikhzadeh A, Nordin M, Axen K. The effects of breath control on intra-abdominal pressure during lifting tasks. Spine (Phila Pa 1976). 2004 Feb 15;29(4):464-9. doi: 10.1097/01.brs.0000092368.90019.d8. PMID 15094544
- [Background] Hoffmeyer-Zlotnik, J. H. (2003). New sampling designs and the quality of data. Developments in applied statistics. Developments in Applied Statistics. Ljubljana: FDV Methodoloski Zvezki, 205-217.
- [Background] Koyuncu A, Kadota JL, Mnyippembe A, Njau PF, Sijali TR, McCoy SI, Bates MN, Harris-Adamson C, Prata N. Heavy Load Carrying and Symptoms of Pelvic Organ Prolapse among Women in Tanzania and Nepal: An Exploratory Study. Int J Environ Res Public Health. 2021 Jan 31;18(3):1279. doi: 10.3390/ijerph18031279. PMID 33572663
- [Background] MacDonald LA, Waters TR, Napolitano PG, Goddard DE, Ryan MA, Nielsen P, Hudock SD. Clinical guidelines for occupational lifting in pregnancy: evidence summary and provisional recommendations. Am J Obstet Gynecol. 2013 Aug;209(2):80-8. doi: 10.1016/j.ajog.2013.02.047. Epub 2013 Mar 1. PMID 23467051
- [Background] Michie S, Richardson M, Johnston M, Abraham C, Francis J, Hardeman W, Eccles MP, Cane J, Wood CE. The behavior change technique taxonomy (v1) of 93 hierarchically clustered techniques: building an international consensus for the reporting of behavior change interventions. Ann Behav Med. 2013 Aug;46(1):81-95. doi: 10.1007/s12160-013-9486-6. PMID 23512568
- [Background] Moss-Morris, R., Weinman, J., Petrie, K., Horne, R., Cameron, L., & Buick, D. (2002). The Revised Illness Perception Questionnaire (IPQ-R). Psychology & Health, 17(1), 1-16. https://doi.org/10.1080/08870440290001494
- [Background] Oxford University Hospitals. (2016). Your recovery after childbirth. Physiotherapy, exercises and advice. NHS Trust.
- [Background] Parden AM, Griffin RL, Hoover K, Ellington DR, Gleason JL, Burgio KL, Richter HE. Prevalence, Awareness, and Understanding of Pelvic Floor Disorders in Adolescent and Young Women. Female Pelvic Med Reconstr Surg. 2016 Sep-Oct;22(5):346-54. doi: 10.1097/SPV.0000000000000287. PMID 27171318
- [Background] Pathak A, Sharma S, Jensen MP. The utility and validity of pain intensity rating scales for use in developing countries. Pain Rep. 2018 Aug 6;3(5):e672. doi: 10.1097/PR9.0000000000000672. eCollection 2018 Sep-Oct. PMID 30534623
- [Background] da Rocha NS, Power MJ, Bushnell DM, Fleck MP. The EUROHIS-QOL 8-item index: comparative psychometric properties to its parent WHOQOL-BREF. Value Health. 2012 May;15(3):449-57. doi: 10.1016/j.jval.2011.11.035. Epub 2012 Feb 9. PMID 22583455
- [Background] Schwarzer, R. (2008). Modeling Health Behavior Change: How to Predict and Modify the Adoption and Maintenance of Health Behaviors. Applied Psychology, 57(1), 1-29. https://doi.org/10.1111/j.1464-0597.2007.00325.x
- [Background] Schwarzer, R., & Schulz. (2013). Berlin Social Support Scales (BSSS) [Data set]. Whitaker Instiutute. https://doi.org/10.13072/midss.490
- [Background] Sharma, R., & Singh, R. (2012). Determination of Safe Carrying Load Limit for Women Carrying Water. Journal of Ergonomics, 02(02). https://doi.org/10.4172/2165-7556.1000103
- [Background] SUVA, the Swiss National Accident Insurance Fund (Ed.). (2019). Gefährdungsermittlung: Heben und Tragen. https://www.suva.ch/de-CH/material/Dokumentationen/beurteilung-der-koerperlichen-belastung-heben-und-tragen-von-lasten-88190d1812918129
- [Background] Tomberge VMJ, Bischof JS, Meierhofer R, Shrestha A, Inauen J. The Physical Burden of Water Carrying and Women's Psychosocial Well-Being: Evidence from Rural Nepal. Int J Environ Res Public Health. 2021 Jul 26;18(15):7908. doi: 10.3390/ijerph18157908. PMID 34360203
- [Background] Tomberge VMJ, Shrestha A, Meierhofer R, Inauen J. Understanding safe water-carrying practices during pregnancy and postpartum: A mixed-methods study in Nepal. Appl Psychol Health Well Being. 2022 May;14(2):691-711. doi: 10.1111/aphw.12325. Epub 2021 Dec 3. PMID 34862740